CLINICAL TRIAL: NCT07300475
Title: Phase 1 Clinical Trial of a Personalized Cancer Immunotherapeutic (PCI) Strategy +/- AB248 (CD8-selective IL-2 Mutein Fusion Protein) in Patients With a New Diagnosis of Triple Negative Breast Cancer Undergoing Neoadjuvant Chemoimmunotherapy
Brief Title: Cancer Immunotherapeutic (PCI) Strategy in Triple Negative Breast Cancer Patients
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-x465
Record Dates: First submitted 2025-12-09; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Triple Negative Breast Cancer
Keywords: Personalized medicine; IL-2; Cancer neoantigen; Personalized cancer immunotherapeutic; Personalized cancer vaccine
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Paclitaxel; Carboplatin; pembrolizumab; Doxorubicin; Cyclophosphamide; poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1: Neoadjuvant SOC KEYNOTE 522 + Adjuvant PCI + Pembrolizumab (Experimental): Patients will be treated with standard of care (SOC) neoadjuvant chemoimmunotherapy according to the KEYNOTE 522 regimen for eight 21-day cycles. Patients will take a 2-week drug holiday from the end of SOC neoadjuvant chemoimmunotherapy to the start of personalized cancer immunotherapeutic (PCI). Patients will receive 5 doses of the PCI + poly-ICLC on Days 1, 4, 8, 15, and 22. Patients will undergo the SOC surgery on Day 29 +/- 5 days. Following surgery, patients will receive 3 additional doses of the PCI + poly-ICLC. Patients will receive 9 doses of SOC adjuvant pembrolizumab on a 21-day cycle. The PCI + poly-ICLC will be given on Days 43, 64, and 85.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Pembrolizumab; Drug: Doxorubicin; Drug: Cyclophosphamide; Biological: Personalized cancer immunotherapeutic (PCI); Other: pVAC tools neoantigen prediction algorithm; Drug: poly-ICLC
- Arm 2: Neoadjuvant SOC KEYNOTE 522 + Adjuvant PCI + Pembrolizumab+AB248 (Experimental): Patients will be treated with standard of care (SOC) neoadjuvant chemoimmunotherapy according to the KEYNOTE 522 regimen for eight 21-day cycles. Patients will take a 2-week drug holiday from the end of SOC neoadjuvant chemoimmunotherapy to the start of personalized cancer immunotherapeutic (PCI). Patients will receive 5 doses of the PCI + poly-ICLC on Days 1, 4, 8, 15, and 22. Patients will also receive 2 doses of AB248 on Days 8 and 22. Patients will undergo the SOC surgery on Day 29 +/- 5 days. Following surgery, patients will receive 3 additional doses of the PCI + poly-ICLC. Patients will receive 9 doses of SOC adjuvant pembrolizumab on a 21-day cycle. The PCI + poly-ICLC will be given on Days 43, 64, and 85.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Pembrolizumab; Drug: Doxorubicin; Drug: Cyclophosphamide; Biological: Personalized cancer immunotherapeutic (PCI); Drug: AB248 (CD8-selective IL-2 mutein fusion protein); Other: pVAC tools neoantigen prediction algorithm; Drug: poly-ICLC

INTERVENTIONS:
Drug: Paclitaxel — As part of the KEYNOTE 522 Regimen, paclitaxel is given intravenously (IV) with a dose 80 mg/m2 on Days 1, 8, and 15 of a 21 day cycle after Step 0 enrollment. Paclitaxel will be given a total of 4 cycles (cycles 1-4).
  Other Names: Onxol; Taxol
Drug: Carboplatin — As part of the KEYNOTE 522 Regimen, carboplatin is given intravenously (IV) with a dose of AUC 1.5 on Days 1, 8, and 15 of a 21 day cycle after Step 0 enrollment. Carboplatin will be given a total of 4 cycles (cycles 1-4).
  Other Names: KYXATA; Paraplatin
Drug: Pembrolizumab — As a part of the KEYNOTE 522 Regimen, pembrolizumab is given intravenously (IV) at a dose of 200 mg on Day 1 of a 21 day cycle after Step 0 enrollment. Pembrolizumab will be given for 8 cycles (cycles 1-8)
  Pembrolizumab will also be given intravenously (IV) at a dose of 200 mg on days 43, 64, and 85 (same as adjuvant PCI) and then 6 additional doses.
  Other Names: Keytruda
Drug: Doxorubicin — As part of the KEYNOTE 522 Regimen, doxorubicin will be given intravenously (IV) at a dose of 60 mg/m2 on Day 1 of a 21 day cycle after Step 0 enrollment. Doxorubicin will be given a total of 4 cycles (cycles 5-8).
  Other Names: Adriamycin; Adriamycin PFS; Adriamycin RDF; Rubex
Drug: Cyclophosphamide — As part of the KEYNOTE 522 Regimen, cyclophosphamide is given intravenously (IV) at a dose of 600 mg/m2 dose on Day 1 of a 21 day cycle after Step 0 enrollment. Cyclophosphamide will be given a total of 4 cycles (cycles 5-8).
  Other Names: Cytoxan; Neosar; Frindovyx
Biological: Personalized cancer immunotherapeutic (PCI) — PCI is given intra-muscular (IM) at 1 mg dose. Each PCI will consists of up to 4 separate injections, with each syringe containing peptides from one of the up to four peptide pools combined with adjuvant poly-ICLC.
  Other Names: CD8-selective IL-2 mutein fusion protein
Drug: AB248 (CD8-selective IL-2 mutein fusion protein) — AB248 is given intravenously (IV) over 30 minutes in 0.15 mg/kg dose. AB248 is given on Days 8 and 22 after Step 1 enrollment.
  Arms: Arm 2: Neoadjuvant SOC KEYNOTE 522 + Adjuvant PCI + Pembrolizumab+AB248
Other: pVAC tools neoantigen prediction algorithm — The pVACtools suite of software tools will be used to identify and prioritize cancer neoantigens based on neoantigen identification algorithms.
Drug: poly-ICLC — Poly-ICLC is mixed with the personalized cancer immunotherapeutic (PCI). The PCI is given intramuscularly (IM) at 1mg dose.

SUMMARY:
This is a phase 1 clinical trial to evaluate the safety, feasibility and immunogenicity of a personalized cancer immunotherapeutic (PCI) strategy with or without CD8-selective IL-2 mutein fusion protein in patients with triple negative breast cancer undergoing neoadjuvant chemoimmunotherapy.

ELIGIBILITY:
Step 0 Inclusion Criteria:

* Newly diagnosed, previously untreated, locally advanced non-metastatic triple negative breast cancer (as defined by the most recent ASCO/CAP guidelines). Permissible staging per AJCC is as follows:

  * T1c, N1-N2
  * T2, N0-N2
  * T3, N0-N2
* At least 18 years of age.
* Adequate tissue available for nucleic acid isolation/PCI design.
* Adequate cardiac function per treating physician and a candidate for the KEYNOTE 522 regimen (or receiving the KEYNOTE 522 regimen for no more than one month).
* Ability to understand and willingness to sign an IRB approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Step 0 Exclusion Criteria:

* Prior or concurrent malignancy whose natural history has the potential to interfere with the safety or efficacy assessment of the investigational regimen. Patients with prior or concurrent malignancy that does NOT meet that definition are eligible for this trial.
* Received prior chemotherapy, targeted therapy, or radiation therapy within the past 12 months.
* Received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent, or with an agent directed to another co-inhibitory T-cell receptor.
* Currently receiving any other investigational agents.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to any agents used in the study.
* Received a live vaccine within 30 days of the first dose of pembrolizumab.
* Active autoimmune disease that has required systemic treatment in the past 2 years.
* Diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of pembrolizumab.
* History of (non-infectious) pneumonitis that required steroids, or current pneumonitis.
* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia. Patients with a known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Function Classification; to be eligible for this trial, patients should be a class 2B or better.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 7 days of study entry.
* Known history of active TB (bacillus tuberculosis).
* Known history of HIV.
* Evidence of chronic hepatitis B virus (HBV) that is detectable on suppressive therapy. Patients with evidence of chronic HBV infection with undetectable HBV viral load on suppressive therapy are eligible. HBV testing not required in the absence of known history of infection.
* History of hepatitis C virus (HCV) infection that has not been cured or that has a detectable viral load. Patients with a history of HCV that has been treated and cured are eligible. Patients with HCV infection who are currently on treatment and have an undetectable HCV viral load are eligible. HCV testing not required in the absence of known history of infection.

Step 1 Inclusion Criteria:

* ECOG performance status ≤ 1 within 10 days of initiation of PCI
* Adequate bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1.0 K/cumm
  * Platelets ≥ 100 K/cumm
  * Hemoglobin ≥ 8.0 g/dL
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine clearance > 30 mL/min by Cockcroft-Gault
* The effects of the PCI on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 6 months after last dose of PCI. Should a woman become pregnant or suspect she is pregnant while participating in this study or should a man suspect he has fathered a child, s/he must inform her treating physician immediately.
* Received at least 4 months of the KEYNOTE 522 regimen.

Step 1 Exclusion Criteria:

* Currently receiving any other investigational agents.
* Pregnant and/or breastfeeding.
* Experiencing ongoing AEs related to the SOC KEYNOTE 522 regimen that have not resolved to < grade 3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2030-01-08 (Estimated); Study Completion 2034-12-09 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) | Step 1 enrollment to 30 days after completion of PCI treatment (estimated time of 115 days)
  Treatment-emergent adverse events (TEAEs) will be assessed via CTCAE v5.
Treatment-related adverse events (TRAEs) | Step 1 enrollment to 30 days after completion of PCI treatment (estimated time of 115 days)
  Treatment-related adverse events (TRAEs) will be assessed via CTCAE v5.
Serious adverse events (SAEs) | Step 1 enrollment to 30 days after completion of PCI treatment (estimated time of 115 days)
  Serious adverse events (SAEs) will be assessed via CTCAE v5.
Feasibility as determined by number of enrolled patients with triple negative breast cancer | Completion of enrollment (1 day for patient)
  Defined as enrolling 24 evaluable patients in 36 months.
Feasibility as determined by time required for PCI design and manufacture | Start of Step 0 Enrollment to PCI completion (estimated time of 24 weeks)
  Defined as completion of design and manufacture within 24 weeks.
Feasibility as determined by rate of successful PCI delivery | Day 1
  Defined as at least 70% of patients receiving at least one dose of PCI.

SECONDARY OUTCOMES:
Immune response as evaluated by ELISPOT analysis. | Step 0 Enrollment to 12 months after PCI completion (estimated time of 18 months and 85 days)
  Samples will be drawn at Step 0 enrollment, day 1, day 15, day 22, day of surgery, day 43, day 64, day 85, and patients randomized to Arm 2 will have an optional draw at Year 1 follow-up.
Recurrence-free survival (RFS) | Step 1 enrollment through completion of follow up (estimated time of 5 years and 85 days)
  Recurrence-free survival is defined as the rate of disease recurrence from Step 1 enrollment until disease recurrence per standard of care assessments or until patient is off study, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: William Gillanders, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://siteman.wustl.edu